CLINICAL TRIAL: NCT05329246
Title: Validation of AI-assisted Clinical Assistant for Effective Management of Cardiovascular Diseases in Primary Health Care: PMcardio-1 Trial
Brief Title: Validation of PMcardio AI-assisted Clinical Assistant in Primary Care
Acronym: PMCARDIO-PT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Powerful Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202106001; CIV-21-09-037810 (Other: Clinical Investigation ID)
Record Dates: First submitted 2021-12-13; First posted 2022-04-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases; Medical Device; Primary Health Care; Electrocardiogram; Dyspnea; Chest Pain; Syncope; Breath Shortness; General Practitioner
Keywords: Cardiovascular Diseases; Medical Device; Primary Health Care; Diagnostic Tool; Artificial Inteligence; A.I. Clinical Assistant; Powerful Medical; PMcardio; Electrocardiogram; ECG; ECG Diagnostic
MeSH Terms: conditions — Cardiovascular Diseases; Dyspnea; Chest Pain; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention Group (Experimental): AI-assisted interpretation of the ECG including the predicted ECG diagnoses, disease-specific anamnestic questions, and patient management recommendations for referral to secondary care, including suggestions for procedures and further diagnostic tests
  Interventions: Device: AI-assisted Clinical Assistant PMcardio
- Control Group (No Intervention): The usual standard of care, with NO AI-based diagnosis or treatment recommendation available.

INTERVENTIONS:
Device: AI-assisted Clinical Assistant PMcardio — PMcardio is an AI-powered clinical assistant in the form of a mobile application empowering non-cardiologist healthcare workers with advanced cardiovascular diagnostic capabilities, recommending patient-specific suggestions for referral and facilitating remote consultations with specialized cardiologists.
  Arms: Experimental Intervention Group

SUMMARY:
This study aimed to analyze and investigate whether the use of the PMcardio clinical assistant leads to a more efficient patient management in primary care and more accessible specialised care compared to usual standards of care and to assess the reliability and safety of the PMcardio smartphone application in the primary care use environment. Additionally, to evaluate time savings and cost saving implications of increased availability of specialised care at the primary care level.

DETAILED DESCRIPTION:
It is a multi-centric, physician-driven, patient-blinded randomized controlled trial of patients presenting to the general practitioner with typical cardiovascular symptoms (specifically, chest pain, syncope, palpitations, or shortness of breath) constituting an electrocardiogram examination. Eligible patients will be enrolled at the participating general practitioner clinics and managed either through the PMcardio platform with AI-assisted diagnostics, patient management recommendations or usual standard of care throughout their initial visit. Enrolled participants will be followed-up through health insurance billing codes and there will be no personal follow-up visits required. The aim of the study is to investigate whether the use of the PMcardio clinical assistant leads to a more efficient patient management in primary care and more accessible specialised care compared to usual standards of care and to assess the reliability and safety of the PMcardio smartphone application in the primary care use environment. Additionally, to assess time savings and cost saving implications of increased availability of specialised care at the primary care level.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 55 years or above.
* Participant is willing and able to give informed consent for participation in the study.
* Presenting to the GP with ANY of the following cardiovascular symptoms: palpitations, chest pain, syncope, shortness of breath.
* Patients insured by Dôvera ZP or Union ZP health insurance providers.

Exclusion Criteria:

* Reason for doing the ECG at the GP clinic is a routine examination or pre-operative assessment.
* Participant does not present with cardiovascular symptoms: palpitations, chest pain, syncope, shortness of breath.
* Participant is already included in the study due to a prior GP visit throughout the trial period (e.g., participant comes for a second visit to GP clinic due to cardiovascular symptoms).
* Patients insured by VšZP health insurance provider
* Female participants who are pregnant, lactating or planning pregnancy during the study.
* Any other significant comorbidity, disease, or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time to first cardiovascular-related consultation | From randomization to enrollment period completion (up to 6 months)
  Time from randomization to the first cardiovascular-related consultation or a follow-up visit at specialized physician in patients, where specialized consultation is indicated based on the general practitioner recommendation after using PMcardio application. The measurement will be assessed from the data received from the health insurance provider.
Time to first cardiovascular-related diagnostic testing | From randomization to to enrollment period completion (up to 6 months)
  Time from randomization to the first cardiovascular-related further diagnostic testing (laboratory parameters, ECG Holter, echocardiography).The measurement will be assessed from the data received from the health insurance provider
Time to first cardiovascular-related hospitalization | From randomization to to enrollment period completion (up to 6 months)
  Time from randomization to the first hospitalization in patients, where hospitalization is indicated, based on the general practitioner recommendation while using PMcardio application. The measurement will be assessed from the data received from the health insurance provider
Time to first cardiovascular-related drug prescription | From randomization to to enrollment period completion (up to 6 months)
  Time from randomization to the first cardiovascular-related drug prescription in patients, where drug prescription is indicated, based on the general practitioner recommendation while using PMcardio application. The measurement will be assessed from the data received from the health insurance provider

SECONDARY OUTCOMES:
Cost-effectiveness ratio and effect on cost savings | 1 year
  Cost-effectiveness ratio and projected effect on cost savings resulting from PMcardio remote specialist consultations measured based on Health Insurance data
Reliability and safety of the PMcardio measured by system up-time | From the very first participants randomization to total follow-up time (up to 6 months)
  The duration of time that the operating system of the application has been working and available in a reliable operating manner.
Reliability and safety of the PMcardio measured by system failures | From the very first participants randomization to total follow-up time (up to 6 months)
  The Number of failures by PMcardio application that caused the system to end abnormally.
General practitioner satisfaction assessed by Client Satisfaction Questionnaire (CSQ-8 scale). | From randomization to study completion (up to 1 year)
  The Client Satisfaction Questionnaire (CSQ-8 scale) measures general satisfaction of participating general practitioners with the functionality of the application at the end of the enrollment period. Possible scores range from 8 to 32, with higher scores indicating higher satisfaction with the application.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hatala, PhD, Principal Investigator — Chief Scientist and Founder
Locations (56):
- Slovakia (56):
  - MUZMED s.r.o., Bardejov
  - MAR-BID s.r.o., Bidovce
  - SIMAMED, s.r.o., Borský Mikuláš
  - SollarMED, s.r.o., Bratislava
  - NÁGEL, s.r.o., Búč
  - MEDIFARMA s.r.o., Dolný Kubín
  - Promedicum, s.r.o., Hanušovce nad Topľou
  - GP Humenné, s.r.o., Humenné
  - LPSo spol. s r.o., Humenné
  - MED - AID s.r.o., Humenné
  - MUDr. Peter Križalkovič, Hurbanovo
  - MUDr. Ildikó Papáčková, Kolárovo
  - BELLIS-med s.r.o., Komárno
  - MEDIKONTAKT, s.r.o., Komárno
  - IRS - Medicínska činnosť s.r.o., Košice
  - MUCOMED s.r.o., Košice
  - MUDr. Ján Telepovský, Košice
  - SANABITUR, s.r.o., Križovany Nad Dudváhom
  - Anahata s.r.o., Lenartovce
  - FONTHIS, s.r.o., Levice
  - MUDr. Mária Schmidtová, s.r.o., Martin
  - Vaša ambulancia, s. r. o., Martin
  - MUDr. Ondrej Gajdoš, Medzev
  - Medic I+H s.r.o., Medzilaborce
  - JANMED, s.r.o., Michalovce
  - Cardio Clinic s.r.o., Moldava nad Bodvou
  - G.Praktik s.r.o., Moldava nad Bodvou
  - HODOSI-MED s.r.o, Moldava nad Bodvou
  - Tamice,s.r.o., Moldava nad Bodvou
  - LEK - NO, s.r.o., Námestovo
  - TOMICI s.r.o., Nesvady
  - Timimed s. r. o., Nitra
  - VERKIAD s.r.o., Nitra
  - VALETUDO s.r.o., Nitrianske Hrnčiarovce
  - RODMED s.r.o., Nové Zámky
  - Duo medical s.r.o., Pezinok
  - PALMED, s.r.o., Podolínec
  - MEDIPRAX s.r.o, Poprad
  - PULSE medicine, s.r.o, Poprad
  - GP - PRAKTIK, s.r.o., Prešov
  - KNG s.r.o., Prešov
  - MDPRAK, s.r.o., Prešov
  - RM - MEDICAL s.r.o., Prievidza
  - CorMedicus s.r.o., Ruskov
  - Jklinik s.r.o, Ružomberok
  - PT Care s.r.o., Spišský Hrušov
  - MUDr. Boris Piteľ, Stakčín
  - MEDICATEK s.r.o., Starý Tekov
  - VINOVA Group s.r.o., Strekov
  - AVK MEDIC, s.r.o., Štúrovo
  - GPII Medical s.r.o., Tekovské Lužany
  - MUDr. Peter MARKO, s.r.o., Veľká Lomnica
  - Resutík s.r.o., Veľký Krtíš
  - MUDr. Viera Čuchranová, Vinne
  - JOMED, spol. s r.o., Vranov nad Topľou
  - MUDr. Orság Juraj, s.r.o., Želiezovce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PMcardio Landing Page — https://www.powerfulmedical.com/